CLINICAL TRIAL: NCT06189183
Title: Adjuvant Hypofractionation Radiotherapy for Thymic Epithelial Tumours After Complete Resection-Single Center Phase II Single Arm Clinical Trial
Brief Title: Adjuvant Hypofractionation Radiotherapy for Thymic Epithelial Tumours After Complete Resection
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cancer Institute and Hospital, Chinese Academy of Medical Sciences (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCC4287
Record Dates: First submitted 2023-12-18; First posted 2024-01-03 (Actual); Last update posted 2024-02-16 (Actual); Status verified 2023-11

CONDITIONS: Thymus Neoplasms
Keywords: Thymus Neoplasms; Adjuvant Radiotherapy
MeSH Terms: conditions — Thymus Neoplasms

STUDY DESIGN:
Intervention Model Description: Adjuvant Hypofractionation Radiotherapy for Thymic Epithelial Tumours After Complete Resection
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adjuvant Hypofractionation Radiotherapy (Experimental): Adjuvant Hypofractionation Radiotherapy for Thymic Epithelial Tumours After Complete Resection
  Interventions: Radiation: Adjuvant Hypofractionation Radiotherapy

INTERVENTIONS:
Radiation: Adjuvant Hypofractionation Radiotherapy — Adjuvant Hypofractionation Radiotherapy for Thymic Epithelial Tumours After Complete Resection

SUMMARY:
The purpose of this study is to evaluate the efficiency and toxicity of adjuvant hypofractionation radiotherapy for thymic epithelial tumours after complete resection.

DETAILED DESCRIPTION:
Adjuvant Radiotherapy(Postoperative radiotherapy) is proposed in stage II and III thymic carcinoma，stage III thymoma，stage IIB B2/B3 thymomas.

Hypofractionation Radiotherapy is used in this study. The purpose of this study is to evaluate the efficiency and toxicity of adjuvant hypofractionation radiotherapy for thymic epithelial tumours after complete resection.

ELIGIBILITY:
Inclusion Criteria:

* Thymoma and Thymic carcinoma confirmed by histology or cytology
* R0 resection (complete resection)
* stage II and III thymic carcinoma，stage III thymoma，stage IIB B2/B3 thymomas.
* Karnofsky performance status(KPS) 80, 90 or 100.
* Having sufficient Pulmonary function, renal function and liver function. Neutrophile granulocyte count>1.5×109 /L, platelet count>80×109 /L, hemoglobin ≥10g/dL.

Exclusion Criteria:

* Prior thoracic radiotherapy.
* Uncontrolled Comorbidities.
* Pregnant or nursing mother.
* Pneumonia

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2023-11-11 (Actual); Primary Completion 2030-12-31 (Estimated); Study Completion 2040-12-31 (Estimated)

PRIMARY OUTCOMES:
Disease Free Survival | 2 years, 5 years
  From the date of resection to the date of disease recurrence or death

SECONDARY OUTCOMES:
Overall Survival | 2 years, 5 years
  From the date of resection to the date of death
RadiotherapyToxicity | 1 years, 2 years, 5 years
  Rate of pneumonitis；Rate of esophagitis；Rate of skin reaction；Rate of myelitis；Rate of heart disease；Rate of vascular toxicity
local recurrence | 2 years, 5 years
  recurrence of tumor bed
Intrathoracic recurrence / pleural metastasis | 2 years, 5 years
  Rate of Intrathoracic recurrence / pleural metastasis
metastasis free survival | 2 years, 5 years
  From the date of resection to the date of metastasis or death

CONTACTS AND LOCATIONS:
Overall Officials: Tao Zhang, Dr., Principal Investigator — National Cancer Center/Cancer Hospital, CAMS
Locations (1):
- National Cancer Center/Cancer Hospital, Chinese Academy of Medical Science and Peking Union Medical College, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No